CLINICAL TRIAL: NCT07030179
Title: The Relationship Between Preoperative Frailty and Postoperative Acute Kidney Injury in Patients Undergoing Non-cardiac Surgery and the Mediating Effect of Intraoperative Blood Pressure: A Prospective Cohort Study
Brief Title: The Relationship Between Preoperative Frailty and Postoperative AKI and the Mediating Effect of Intraoperative BP
Status: Recruiting | Type: Observational
Sponsor: Lanyue Zhu (Other)
Responsible Party: Sponsor-Investigator, Lanyue Zhu, Attending Doctor, Zhongda Hospital
Organization: Zhongda Hospital (Other)
Other Study IDs: 2025ZDSYLL201-P01
Record Dates: First submitted 2025-06-07; First posted 2025-06-22 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-06

CONDITIONS: Postoperative Acute Kidney Injury; Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Frail group: We chose the Fried Phenotypic Assessment Scale to evaluate the frailty status of the patients. The Fried Frailty Assessment Scale holds that frailty is a syndrome composed of five phenotypes: shrinking, weakness, exhaustion, low physical activity, and slowness. Meeting three or more of these phenotypes indicates a frailty status.
  Interventions: Other: Frailty status
- Non-frail group: We used the Fried assessment scale to evaluate the frailty status of patients. Patients who met two or fewer indicators were evaluated as having a non-frailty status.

INTERVENTIONS:
Other: Frailty status — This was an observational study with no intervention measures. The exposure factor was the frailty status of the patients.
  Groups: Frail group

SUMMARY:
The primary objectives of study is to compare the difference in the incidence of postoperative AKI between frail and non-frail patients. The secondary objectives of study was to compare the differences in intraoperative blood pressure fluctuations, the incidence and duration of intraoperative hypotension, postoperative complications, length of hospital stay and hospitalization expenses between frail and non-frail patients, and use mediating effect analysis to examine the magnitude of the effect of intraoperative blood pressure on postoperative acute kidney injury caused by frailty.

DETAILED DESCRIPTION:
This study is a single-center prospective cohort study. It is expected to include patients who meet the inclusion and exclusion criteria from July 2025 to February 2026. The demographic characteristics, laboratory indicators, preoperative comorbidities of the patients will be recorded and frailty assessment will be conducted within one week before the operation. The patients were divided into the frail group and the non-frail group. Record the surgery-related information of the patient on the day of the operation. During the operation, vital signs such as the patient's blood pressure and heart rate were routinely detected. The anesthesiologist adopted an experience-guided anesthesia management approach, and the doctor in charge of anesthesia management was also unaware of the patient's frailty status. Record the indicators such as the dosage of anesthetic drugs during the operation, the duration of surgical anesthesia, the use of vasoactive drugs and the fluid intake and output of the patients. The incidence of AKI, the incidence of in-hospital complications, the length of hospital stay and the hospitalization costs of the patients were recorded after the operation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or above
* Undergo non-cardiac surgery

Exclusion Criteria:

* At least one measurement of serum creatinine (SCr) was not conducted before and after the operation
* End-stage renal disease (ESRD) that has received dialysis within the past year
* Baseline SCr ≥ 4.5 mg/dl (because the clinical criteria for AKI based on elevated SCr may not be applicable to these patients)
* Acute kidney injury occurred within 7 days before the operation
* No frailty assessment was conducted
* The operation time is less than 2 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent non-cardiac surgery at Zhongda Hospital Southeast University.
Sampling Method: Non-Probability Sample
Enrollment: 515 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative acute kidney injury | Within one week after the operation

SECONDARY OUTCOMES:
Intraoperative blood pressure | During the operation
Postoperative complications | Perioperative period
Hospital stays | Perioperative period
Hospitalization costs | Perioperative period

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital Southeast University, Nanjing, Jiangsu, China